CLINICAL TRIAL: NCT01723956
Title: Validation of Implementation of Cervical Dysplasia Treatment Modalities in HIV-Seropositive Women
Acronym: VICAR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Cynthia S Firnhaber, Associate Professor of Medicine, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZA.09.0265
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-08

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cervical Dysplasia; Cin 2; Cin 3; HIV positive women; South Africa
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm B (Active Comparator): LEEP treatment of CIN 2/3 cervical lesion in HIV positive women (standard of Care)
  Interventions: Procedure: LEEP
- Arm A (Experimental): Cryotherapy treatment of CIN 2/3 cervical lesions
  Interventions: Procedure: Cryotherapy

INTERVENTIONS:
Procedure: Cryotherapy — This is involves freezing the lesions with a cryo gun using Nitrous Oxide for 3 minutes-- wait 5 minutes and then refreezing for 3 more minutes. This procedure uses the Wallach cryogun
  Other Names: This is a study using Freezing with a cryogun
  Arms: Arm A
Procedure: LEEP — The cervix is anaesthetized with lidocaine and then a electric loop is applied to the cervical lesion which is cut with one pass. The LEEP machine used is the automatic Finesse Machine.
  Other Names: Loop Electric Excision Procedure
  Arms: Arm B

SUMMARY:
To compare the efficacy of cryotherapy and large loop excision of the transformation zone (LLETZ) procedures for the treatment of high-grade cervical intra-epithelial neoplasia (CIN2/3) among HIV-seropositive women by follow-up VIA, cytology and Human Papillomavirus.

Hypothesis: LEEP will be more effective than cryotherapy in removing CIN 2/3 lesions in HIV positive women in South Africa

DETAILED DESCRIPTION:
Cervical cancer is the most common cancer in HIV positive women. This is due to immunosuppression and lack of organized and effective screening and treatment programs in Africa. Other screening and treatment modalities need to be evaluated in resource limited countries as there is not capacity in most of these countries to implement a cytology/histology based program. The treatment modality of cryotherapy is easy to train and perform and can be done by a nurse. LEEP requires significant training usually doctors and skills in administering local anaesthetic. This study compares the two modalities of cryotherapy vs LEEP in a randomized controlled study in HIV positive women in South Africa.

A. PRIMARY AIMS (S.A.):

1. To compare the efficacy of cryotherapy and large loop excision of the transformation zone (LLETZ) procedures for the treatment of high-grade cervical intra-epithelial neoplasia (CIN2/3) among HIV-seropositive women by follow-up VIA, cytology and HPV.
2. To determine the utility of subsequent HPV DNA testing as a marker of effective treatment following the treatment of CIN 2/3 among HIV-seropositive women.
3. To compare the safety of cryotherapy versus LLETZ in HIV seropositive women.

SECONDARY AIMS:

1. To describe HIV disease status (CD4, HIV viral load), demographics, and sexual behavior in each treatment arm (LLETZ and cryotherapy) in HIV seropositive women.

3. To determine the cervical disease recurrence rates with cryotherapy and LLETZ.

4. To evaluate the relationship between HIV status, demographics, HPV, and sexual behavior with the clearance of cervical disease at the ectocervical and endocervical margins in HIV seropositive women.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-65 years of age
* Not menstruating (if menstruating, the patient can be screened at another date)
* Able to sign consent
* Able to follow the study protocol
* HIV positive (by two different criteria; either 2 different rapid HPV tests of different manufacturers, a HIV viral load ≥5,000,ELISA, Western blot documented in VICAR 1)
* Participant with histology-proven CIN 2 or 3 disease

Exclusion Criteria:

* Pregnant
* Clinically active sexually transmitted disease determined by clinical history and/or physical exam (may participate after adequate treatment by syndromic treatment management)
* Known and previous treatment for high grade squamouse intraepithelial lesion by any method (cryotherapy, LLETZ or cone biopsy)
* Previous hysterectomy with removal of the cervix
* Significant medical illness/mental illness that the investigator feels would prevent the participant from complying with the protocol or place the participant at medical risk
* Cervical dysplastic lesions that are not appropriate for cryotherapy, defined as the following:

  1. Lesion is greater than ≥75% cervix
  2. Lesion entering into the cervical canal and the complete lesion cannot be visualized
  3. Presence of abnormal vasculature
  4. Lesion bigger that the cryotherapy probe

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2010-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Compare efficacy of cryotherapy and LEEP | 1 year
  To compare the efficacy of cryotherapy and large loop excision of the transformation zone (LLETZ) procedures for the treatment of high-grade cervical intra-epithelial neoplasia (CIN2/3) among HIV-seropositive women by follow-up VIA, cytology and HPV.

SECONDARY OUTCOMES:
The ability to use Human Papillomavirus as the measure of treatment success | 1 year
  To determine the utility of subsequent HPV DNA testing as a marker of effective treatment following the treatment of CIN 2/3 among HIV-seropositive women.
To compare the safety of cryotherapy versus LLETZ in HIV seropositive women | 1 month, 6 months and 12 months
  To compare the safety of cryotherapy versus LLETZ in HIV seropositive women by evaluating adverse events as measured by the Division of AIDS toxicity table 2004 (revised August 2010)
Describe factors associated with successful treatment of CIN 2/3 | 1 year
  To describe HIV disease status (CD4, HIV viral load), demographics, tissue margins and sexual behavior in each treatment arm (LLETZ and cryotherapy) in HIV seropositive women.
To determine the cervical disease recurrence rates with cryotherapy and LLETZ. | 6 months and 12 months
  To determine the cervical disease recurrence rates with cryotherapy and LLETZ at 6 months and 12 months by colposcopy

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia S Firnhaber, MD, Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- Helen Joseph Hospital, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Derived] Smith JS, Sanusi B, Swarts A, Faesen M, Levin S, Goeieman B, Ramotshela S, Rakhombe N, Williamson AL, Michelow P, Omar T, Hudgens MG, Firnhaber C. A randomized clinical trial comparing cervical dysplasia treatment with cryotherapy vs loop electrosurgical excision procedure in HIV-seropositive women from Johannesburg, South Africa. Am J Obstet Gynecol. 2017 Aug;217(2):183.e1-183.e11. doi: 10.1016/j.ajog.2017.03.022. Epub 2017 Mar 31. PMID 28366730